CLINICAL TRIAL: NCT04839432
Title: Effect of 4% Albumin Prime Solution for Cardiopulmonary Bypass on Postoperative Pulmonary Complications In Patients Undergoing Pulmonary Endarterectomy: A Propensity-adjusted Analysis
Brief Title: Crystalloids vs Albumin Prime Solution and Postoperative Pulmonary Complications
Acronym: ALBUTEP
Status: Completed | Type: Observational
Sponsor: Erasme University Hospital (Other)
Responsible Party: Principal Investigator, Alexandre Joosten, MD PhD, Study Director, Erasme University Hospital
Other Study IDs: IRB 00012157
Record Dates: First submitted 2021-04-07; First posted 2021-04-09 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Crystalloids group: Patients had only a balanced crystalloid solution in the priming of the cardiopulmonary bypass (pre interventional group)
- albumin group: Patients had only a 4% albumin solution in addtion to a very low volume of a balanced crystalloid solution in the priming of the cardiopulmonary bypass (post interventional group)
  Interventions: Behavioral: implementation of albumin solution in the priming of the cardiopulmonary bypass machine

INTERVENTIONS:
Behavioral: implementation of albumin solution in the priming of the cardiopulmonary bypass machine — In March 2019, the investigators initiated a new priming fluid policy strategy aiming at replacing our traditional pure crystalloid fluid administration for an albumin one in order to decrease the relatively high-rate of observed pulmonary complications
  Groups: albumin group

SUMMARY:
In 2019, the investigators initiated a new priming fluid therapy strategy in the cardiopulmonary bypass (CPB) machine for patients undergoing pulmonary endarterectomy surgery. It consisted in a transition from a "pure" primarly balanced crystalloid priming fluid strategy to a 4% human albumin priming fluid-strategy in addition to a low volume of balanced crystalloid solution. The rationale was the theoritical assumption that albumin leads to better intravascular volume expansion compared to crystalloid and therefore could reduce overall volume requirement during surgery and consequently potentially decrease the incidence of postoperative pulmonary complications. The objective of this propensity-matched study was to evaluate the effectiveness of this intervention

DETAILED DESCRIPTION:
Intravenous fluid is usually needed (and sometime in important amount) to increase intravascular volume during cardiac surgery and to prime the cardiopulmonary bypass (CPB) circuit. In this context, albumin has been frequently used as the ideal fluid choice. Although albumin has the disadvantage to be much more expensive than crystalloids and not to be free from immunological reactions, this solution provides a more sustained volume effect that a similar volume of crystalloid which may result in smaller volumes of resuscitation fluid being administered. It also better preserves the on-bypass oncotic pressure and reduce extravascular lung water. These considerations are important especially during pulmonary thromboendarterectomy surgery (PTE), a high-risk procedure which aims to resect thromboembolic material. Reperfusion lung injury (RLI) and/or acute respiratory distress syndrome (ARDS), are the most encountered postoperative pulmonary complications and are significant risks factors of morbi-mortality. As data suggest that RLI and ARDS are high-permeability phenomenon, cautious is required to avoid fluid accumulation/overload during this complex procedure. In addition, this surgical procedure has a relatively high CPB duration which can induce a systemic inflammatory response syndrome, damage the endothelial glycocalyx and vascular barrier where crystalloids may extravagates and accumulates in the lungs. On the contrary, albumin solution used during the priming of CPB can favorably preserve oncotic pressure, have a protective effect on endothelial glycocalyx and better maintain vascular barrier competence, preventing interstitial edema and potential pulmonary complications.

In March 2019, the investigators initiated a new priming fluid policy strategy aiming at replacing our traditional pure crystalloid fluid administration for an albumin one in order to decrease the relatively high-rate of pulmonary complications observed in the investigators patients.

The objective of this propensity-matched study was to evaluate the effectiveness of this intervention

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients undergoing pulmonary endarterectomy surgery

Exclusion Criteria:

* Patients with important missing data
* Patients undergoing combined surgery
* Patients undergoing an emergency pulmonary endarterectomy surgery

Ages: 14 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients undergoing pulmonary endarterectomy surgery from 2018 to 2019 ( a two years study period)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
pulmonary complications | postoperative day 7
  a composite of two pulmonary complications ( reperfusion lung syndrome and/or acute respiratory distress syndrome)

CONTACTS AND LOCATIONS:
Overall Officials: Amelie Delaporte, MD, Principal Investigator — Marie lannelongue
Locations (1):
- Marie lannelongue, Le Plessis-Robinson, Paris, France